CLINICAL TRIAL: NCT05757245
Title: A Phase 1 Open Label Study Evaluating the Safety and Efficacy of Gene Therapy in Subjects With Transfusion-dependent α-Thalassemia by Transplantation of Autologous CD34+ Cells Transduced Ex Vivo With a Lentiviral Vector (GMCN-508A Drug Product)
Brief Title: A Study Evaluating the Safety and Efficacy of the GMCN-508A Drug Product in Transfusion-dependent α-Thalassemia Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Genmedicn Biopharma Ltd. (Unknown)
Responsible Party: Principal Investigator, Yongrong Lai, MD, Director of Hematology Department of First Affiliated Hospital of Guangxi Medical University, First Affiliated Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMCN-508A-01
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Transfusion-dependent α-Thalassemia
Keywords: GMCN-508A; gene therapy; Transfusion-dependent α-Thalassemia; Human Hematopoietic Stem Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMCN-508A (Experimental): GMCN-508A infusion
  Interventions: Genetic: GMCN-508A Drug Product

INTERVENTIONS:
Genetic: GMCN-508A Drug Product — Transplant of autologous hematopoietic stem and progenitor cells transduced with GMCN-508A lentiviral vector.

SUMMARY:
This is a non-randomized, open label, single-site, single-dose, phase 1 study in up to 5 participants (between 5 and 35 years of age, inclusive) with Transfusion-dependent α-thalassemia. The study will evaluate the safety and efficacy of autologous hematopoietic stem cell transplantation (HSCT) using GMCN-508A Drug Product [autologous CD34+ hematopoietic stem cells transduced with GMCN-508A lentiviral vector encoding the human α-globin gene].

DETAILED DESCRIPTION:
Subject participation for this study will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. The subject himself/herself or one legal guardian/agent of the subject is required to fully understand the study and voluntarily sign a written informed consent.
2. Ages 5 to 35, no gender limitation.
3. The clinical diagnosis of Transfusion-dependent α-Thalassemia.Transfusion dependence was defined as ≥6 Units of transfusions of pRBCs for the prior 24 weeks without >56 days of non-transfusion.
4. Karnofsky Level of Performance (KPS) score or Lansky Level of Performance (LPS) score ≥70.
5. Subjects were determined to undergo autologous hematopoietic stem cell transplantation and conditioning procedure by the principle investigator.
6. Subjects were willing to comply with the protocol.
7. Fertile Subjects are willing to take effective contraceptive measures during the study.

Exclusion Criteria:

1. Diagnosed with mild α-thalassemia, Hb Bart's edema, ATRx α-thalassemia, hemoglobin S/β-thalassemia, myelodysplastic subtype anemia, or with HbE homozygous β gene mutation, or with any type of β-thalassemia Thalassemia.
2. Uncorreted Bleeding disorders with frequent bleeding (eg, menorrhagia, epistaxis, coagulation disorders).
3. Bacterial, fungal, parasitic or viral infection as determined by the investigator to be clinically significant.
4. Presence of severe iron overload.
5. Any prior or current malignancy, myeloproliferative disorders or immunodeficiency disorders.
6. Any major medical disease, laboratory test abnormality or mental illness that would render the participant ineligible for the study.
7. Immediate family member with a known Familial Cancer Syndrome.
8. Prior receipt of gene therapy, allogeneic bone marrow transplantation or allogeneic hematopoietic stem cell transplantation.
9. Participation in another clinical study with an investigational drug 3 months prior to Screening.
10. Pregnancy, plan to be pregnant during study or breastfeeding in a postpartum female.
11. Known hypersensitivity to any ingredients or excipients of the test drug.
12. Eligible for allogeneic bone marrow transplantation or allogeneic hematopoietic stem cell transplantation with a known and available donor.
13. Any other condition that would render the participant ineligible for the study, as determined by the investigator.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-05-08 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved Transfusion Independence (TI) | From time of drug product infusion up to 24 months
  TI was defined as a weighted average hemoglobin (Hb) >= 9 g/dL without any packed red blood cells (pRBC) transfusions for a continuous period of >=12 months at any time during the study after GMCN-508A Drug Product infusion. Percentage of participants who achieved TI from time of drug product infusion up to 24 months was reported.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved Transfusion Independence (TI) at Month 24 | Month 24
  TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after GMCN-508A Drug Product infusion.
Duration of Transfusion Independence (TI) | From time of drug product infusion up to 24 months
  TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after GMCN-508A Drug Product infusion. Time period of TI will start when participants achieve a Hb >= 9 g/dL with no transfusions in the preceding 60 days. Duration of TI was calculated as the time from the start of TI (i.e. first Hb >= 9 g/dL with no transfusions in the preceding 60 days) up to the last available Hb at which the TI criteria are still met.
Time From GMCN-508A Drug Product Infusion to Achieving Transfusion Independence (TI) | From time of drug product infusion up to 24 months
  TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after GMCN-508A Drug Product infusion. Time from drug product infusion to initial achievement of TI was calculated as the time from drug product infusion to the first Hb at which a participant can be declared as TI.
Weighted Average Hemoglobin (Hb) During Period of Transfusion Independence (TI) | From time of drug product infusion up to 24 months
  The weighted average Hb is an average area under the curve during the period of TI, from the start of TI when the Hb is first >= 9 g/dL with no transfusions in the preceding 60 days to the last available Hb at which the TI criteria are still met.
Annualized Number of pRBC Transfusions | From 12 to 24 months post drug product infusion
  Annualized number of pRBC transfusions from 12 months post-drug product infusion through Month 24 compared to the annualized number of transfusions during the 24 months prior to enrollment.
Annualized Volume of pRBC Transfusions | From 12 to 24 months post drug product infusion
  Annualized volume of pRBC transfusions from 12 months post-drug product infusion through Month 24 compared to the annualized volume of transfusions during the 24 months prior to enrollment.
Proportion of Participants Who Have Not Received Chelation Therapy for At Least 6 Months Following Drug Product Infusion. | From 6 to 24 months
Change From Baseline in liver Iron Content by Magnetic Resonance Imaging (MRI) | Baseline, Month 12 and 24
Change From Baseline in Cardiac T2* on MRI | Baseline, Month 12 and 24
Change From Baseline in Serum Ferritin | Baseline, Month 12 and 24
Time to Neutrophil Engraftment | From time of drug product infusion up to 24 months
  Time to neutrophil engraftment was defined as the time to the first of 3 consecutive absolute neutrophil count (ANC) >= 0.5 × 10^9/L obtained on different days after a post-transplant value of < 0.5 × 10^9/L. The Day of neutrophil engraftment is the first day of the 3 consecutive measurements, where Day 0 is the day of drug product infusion.
Proportion of Participants With Successful Platelet Engraftment | From time of drug product infusion up to 24 months
  Platelet engraftment was defined as achieving 3 consecutive platelet values >= 20 × 10^9/L on different days after a post-transplant value of < 20 × 10^9/L, while no platelet transfusions administered for 7 days immediately preceding and during the evaluation period.
Time to Platelet Engraftment | From time of drug product infusion up to 24 months
  Platelet engraftment was defined as achieving 3 consecutive platelet values >= 20 × 10^9/L on different days after a post-transplant value of < 20 × 10^9/L, while no platelet transfusions administered for 7 days immediately preceding and during the evaluation period.
Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale (GCS) Score | Baseline, Month 12 and 24
  PedsQL GCS is designed to measure health-related quality of life in pediatric participants and adolescents (2 to 18 years of age). It encompasses 4 dimensions of functioning (physical [8 items], emotional [5 items], social [5 items], school [3 items]). Age groups: Toddler (2-4 years), Young pediatric (5-7 years), Pediatric (8-12 years), and Teens (13-18 years). Depending on the participant's age, the questionnaire may be completed by parent/caregiver as appropriate. For the Toddler group, the PedsQL GCS consist of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consist of 23 items, with a 3-point Likert scale (0, 2, 4) for the young pediatric, and a 5-point Likert scale for the pediatric and teens groups. Scores are transformed on a scale from 0 to 100 where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Change From Baseline in Short Form-36 Health Survey (SF-36) | Baseline, Month 12 and 24
  SF-36 is a generic quality-of-life instrument that had been widely used to assess HRQL of participants. Generic instruments were used in general populations to assess a wide range of domains applicable to a variety of health states, conditions, and diseases. The SF-36 consisted of 36 items that were aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of the time to 5=none of the time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of the time to 5=all of the time], social functioning [1=all of the time: to 5=none of the time], role emotional [1=all of the time to 5=none of the time] and mental health [1=all of the time to 5=none of the time]), with scores ranged from 0 to 100. Higher scores indicating better HRQL.
Proportion of Participants With Successful Neutrophil Engraftment | From time of drug product infusion up to 24 months
  Neutrophil engraftment was defined as achieving 3 consecutive absolute neutrophil count (ANC) >= 0.5 × 10^9/L on different days after a post-transplant value of < 0.5 × 10^9/L within 42 days after drug product infusion.
Transplant-related Mortality | Through 100 and 365 days post GMCN-508A Drug Product infusion
  Transplant-related mortality was determined by the investigator (any deaths considered related to the transplant.)
Proportions of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From signing of informed consent to 24 months after the drug product infusion
  An AE was defined as any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE was any AE, occurring at any dose and regardless of causality that: results in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect.
Overall Survival | From time of drug product infusion up to 24 months
  Overall survival was defined as time from date of GMCN-508A Drug Product infusion (Day 0) to date of death. Overall survival was censored at the date of last visit if the participant was still alive. Percentage of participants who survived throughout the study were reported.
Incidence of acute and/or chronic graft-versus-host disease (GVHD) | From time of drug product infusion up to 24 months
  acute and/or chronic graft-versus-host disease (GVHD) was determined by the investigator.
Percentage of Participants Detected With Replication-competent Lentivirus (RCL) | From time of drug product infusion up to 24 months
Percentage of Participants with occurrence of malignant disease | From time of drug product infusion up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of guangxi medical university, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No